CLINICAL TRIAL: NCT04615052
Title: Home-based Exercise Training in COVID-19 Survivors: a Randomized Controlled Trial
Brief Title: Home-based Exercise in COVID-19 Survivors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Bruno Gualano, Professor, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 4.342.082
Record Dates: First submitted 2020-10-29; First posted 2020-11-04 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2022-06

CONDITIONS: Covid19; SARS (Severe Acute Respiratory Syndrome); SARS-CoV Infection
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — Exercise

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise group (Experimental)
  Interventions: Other: Exercise training
- Control group (No Intervention): The control group will receive all regular medical care and advice on healthy lifestyle including the promotion of recommended physical activity levels.

INTERVENTIONS:
Other: Exercise training — A 16 weeks parallel-group randomised controlled trial will be performed, in which covid-19 survivors patients will complete a telemonitored home-based exercise training program, 3 times per week. The training program will involve strength, aerobic, balance and flexibility exercises.
  Arms: Exercise group

SUMMARY:
The physical inactivity promoted by the patient's hospitalization, including those infected with the coronavirus, can lead to an important health impairment, including atrophy and loss of muscle function. Thus, a prospective study will be conducted to assess the effect of a home-based exercise training program on health outcomes and quality of life in COVID-19 survivors.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with COVID-19
* Positive RT-PCR test and/or serology assay to detect IgG against SARS-CoV-2 in addition to acute symptomatology compatible with the disease
* Admitted in intensive care unit

Exclusion Criteria:

* Cardiovascular disease
* Resting dyspnea
* Acute pulmonary embolism or pulmonary infarction
* Deep venous thromboembolism
* Uncontrolled visual or vestibular disorders
* Pregnancy
* Uncontrolled resting tachycardia
* Uncontrolled hypertension
* Uncontrolled Type II diabetes
* Acute infections
* Neurological disorders
* Patients with chronic kidney disease who are in need of hemodialysis
* Recent malignant neoplasm (<5 years)
* Autoimmune diseases
* Complex ventricular arrhythmias, atrial fibrillation or complete heart block
* Transplant patients
* Any physical disabilities that could hamper physical testing and exercise program

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2020-09-26 (Actual); Primary Completion 2022-09-30 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline on quality of life assessed by the SF-36 health survey questionnaire at 16 weeks. | Baseline and 16 weeks.
  Higher score means better outcome.

SECONDARY OUTCOMES:
Change from baseline on fatigue evaluated by the fatigue severity scale at 16 weeks. | Baseline and 16 weeks.
  Higher score means worse outcome.
Change from baseline on lipid profile at 16 weeks. | Baseline and 16 weeks.
  Total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides
Change from baseline on insulin sensitivity at 16 weeks. | Baseline and 16 weeks.
  Fasting serum concentrations of glucose and insulin.
Change from baseline on inflammatory cytokine IL-1 at 16 weeks. | Baseline and 16 weeks.
Change from baseline on inflammatory cytokine IL-1ra at 16 weeks. | Baseline and 16 weeks.
Change from baseline on inflammatory cytokine IL-6 at 16 weeks. | Baseline and 16 weeks.
Change from baseline on inflammatory cytokine IL-10 at 16 weeks. | Baseline and 16 weeks.
Change from baseline on inflammatory cytokine TNF-alpha at 16 weeks. | Baseline and 16 weeks.
Change from baseline on C-reactive Protein at 16 weeks. | Baseline and 16 weeks.
Change from baseline on Creatine Kinase at 16 weeks. | Baseline and 16 weeks.
Change from baseline on cardiopulmonary fitness assessed by a maximal exercise test at 16 weeks. | Baseline and 16 weeks.
Change from baseline on lean body mass assessed by Dual-energy absorptiometry at 16 weeks. | Baseline and 16 weeks.
Change from baseline body fat assessed by Dual-energy absorptiometry at 16 weeks. | Baseline and 16 weeks.
Change from baseline on waist circumference at 16 weeks. | Baseline and 16 weeks.
Change from baseline on hip circumference at 16 weeks. | Baseline and 16 weeks.
Change from baseline on body weight at 16 weeks. | Baseline and 16 weeks.
Change from baseline on muscular strength assessed by handgrip test at 16 weeks. | Baseline and 16 weeks.
Change from baseline on muscular function assessed by Timed-Stand Test at 16 weesks. | Baseline and 16 weeks.
Change from baseline on muscular function assessed by Timed-Up and Go Test at 16 weeks. | Baseline and 16 weeks.
Change from baseline on anxiety symptoms assessed by Back Scale at 16 weeks. | Baseline and 16 weeks.
  Higher score means worse outcome.
Change from baseline on depression symptoms assessed by Back Scale at 16 weeks. | Baseline and 16 weeks.
  Higher score means worse outcome.
Change from baseline on functional status assessed by Post-COVID-19 Functional Status (PCFS) Scale at 16 weeks. | Baseline and 16 weeks.
  Higher score means worse outcome.
Change from baseline on physical activity levels evaluated by the International Physical Activity Questionnaire at 16 weeks. | Baseline and 16 weeks.
Change from baseline on resting blood pressure assessed by an automated device at 16 weeks. | Baseline and 16 weeks.
Change from baseline on fatigue assessed by Chalder scale at 16 weeks. | Baseline and 16 weeks.
  Higher score means worse outcome.
Change from baseline on heart rate variability assessed by heart rate monitor at 16 weeks. | Baseline and 16 weeks.
Change from baseline on inspiratory muscular strength assessed by power breathe at 16 weeks. | Baseline and 16 weeks.
Change from baseline on quality of life assessed by the SF-36 health survey questionnaire at one year. | Baseline and one year.
  Higher score means better outcome.
Change from baseline on fatigue evaluated by the fatigue severity scale at one year. | Baseline and one year.
  Higher score means worse outcome.
Change from baseline on fatigue assessed by Chalder scale at one year. | Baseline and one year.
  Higher score means worse outcome.
Change from baseline on functional status assessed by Post-COVID-19 Functional Status (PCFS) Scale at one year. | Baseline and one year.
  Higher score means worse outcome.
Change from baseline on muscular function assessed by Timed-Up and Go Test at one year. | Baseline and one year.
Change from baseline on muscular function assessed by Timed-Stand Test at one year. | Baseline and one year.
Change from baseline on muscular strength assessed by handgrip test at one year. | Baseline and one year.
Change from baseline on cardiopulmonary fitness assessed by a maximal exercise test at one year. | Baseline and one year.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Sao Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Longobardi I, Goessler K, de Oliveira Junior GN, Prado DMLD, Santos JVP, Meletti MM, de Andrade DCO, Gil S, Boza JASO, Lima FR, Gualano B, Roschel H. Effects of a 16-week home-based exercise training programme on health-related quality of life, functional capacity, and persistent symptoms in survivors of severe/critical COVID-19: a randomised controlled trial. Br J Sports Med. 2023 Oct;57(20):1295-1303. doi: 10.1136/bjsports-2022-106681. Epub 2023 May 10. PMID 37164620